CLINICAL TRIAL: NCT04535271
Title: TAGGED: A Phase 2 Study Using Low Dose/Metronomic Trabectedin, Gemcitabine, and Dacarbazine as 2nd/3rd/4th Line Therapy for Advanced Soft Tissue Sarcoma
Brief Title: Metronomic Trabectedin, Gemcitabine, and Dacarbazine for Soft Tissue Sarcoma
Acronym: TAGGED
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sarcoma Oncology Research Center, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOC-2101
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Leiomyosarcoma
MeSH Terms: conditions — Leiomyosarcoma | interventions — Trabectedin; Gemcitabine; Dacarbazine

STUDY DESIGN:
Intervention Model Description: This is an open label phase 2 study using metronomic doses of trabectedin, gemcitabine and dacarbazine given intravenously.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Trabectedin 24 h CIV 0.5 mg/m2 D1 and D8 Gemcitabine i.v. 250 mg/m2 D1 and D8 Dacarbazine i.v. 250 mg/m2 D1 and D8
  Interventions: Drug: Trabectedin

INTERVENTIONS:
Drug: Trabectedin — This is an open label phase 2 study using metronomic doses of trabectedin, gemcitabine and dacarbazine given intravenously.
  Other Names: Gemcitabine; Dacarbazine

SUMMARY:
This is an open label phase 2 study using metronomic doses of trabectedin, gemcitabine and dacarbazine given intravenously.

DETAILED DESCRIPTION:
This is an open label phase 2 study using metronomic doses of trabectedin, gemcitabine and dacarbazine given intravenously.

A total of 80 patients will receive trabectedin 0.5 mg/m2 as 24 hour continuous intravenous infusion (CIV) on D1 and D8, gemcitabine 200 mg/m2 i.v. on D1 and D8, and dacarbazine 200 mg/m2 i.v. on D1 and D8 (see product information; www.accessdata.fda.gov). Treatment cycles are given every 3 weeks. Patients in this study may continue treatment until significant disease progression or unacceptable toxicity occurs up to one year of therapy. Patients who withdraw or do not complete the first 2 treatment cycles and first follow up CT scan/MRI will be replaced.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female ≥ 18 years of age
* Pathologically confirmed diagnosis of locally advanced, unresectable or metastatic leiomyosarcoma
* Previously treated patient with measurable disease by RECIST v1.1
* ECOG performance status ≤ 2
* Life expectancy of at least 3 months
* Acceptable liver function: Bilirubin < 1.5 times upper limit of normal (ULN; except subjects with Gilbert Syndrome who must have a total bilirubin level < 3.0 ULN); AST (SGOT), ALT (SGPT) and alk phos < 2.5 x ULN (< 5 x ULN if liver metastases present)
* Acceptable renal function: Creatinine < 1.5 times ULN and creatinine clearance > 60 ml/min using the Crockroft-Gault formula
* Acceptable hematologic status: ANC >1000 cells/μL; Platelet count >100,000/μL; Hemoglobin > 9.0 g/dL
* INR and PT < 1.5 ULN unless taking anti-coagulation, in which case PT, INR and aPTT must be within therapeutic range of intended use of anticoagulants
* Ability to understand the purposes and risks of the study and has signed and dated a written informed consent form approved by the Investigator's IRB/Ethics Committee
* Willingness to comply with all study procedures and availability for the duration of the study
* All women of childbearing potential must have a negative urine or serum pregnancy test within 72 hours of enrollment. If urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required; all subjects must agree to use highly effective means of contraception (surgical sterilization or the use of barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) with their partner from entry into the study through 5 months for women and 7 months for men after the last dose.

Exclusion Criteria:

* Currently receiving treatment with another investigational device or drug study, or <14 days since ending treatment with another investigational device or drug study(s).
* Subject has known sensitivity to trabectedin, gemcitabine or dacarbazine.
* Female subject is pregnant or breast-feeding or planning to become pregnant during study treatment and through 3 months after the last dose of trabectedin, gemcitabine or dacarbazine.
* Female subject of childbearing potential who is unwilling to use acceptable method(s) of effective contraception during study treatment and through 3 months after the last dose of trabectedin, gemcitabine or dacarbazine.
* Sexually active subjects and their partners unwilling to use male or female latex condom

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 12 months
  Progression free survival up to disease progression or death from any cause

SECONDARY OUTCOMES:
Overall Response | 6 weeks
  Best overall response (BOR) and duration of response (DOR) by RECIST v1.1 via CT scan or MRI
Adverse Event | 12 months
  Incidence of treatment-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Sant P Chawla, MD, Principal Investigator — Sarcoma Oncology Research Center, LLC
Locations (1):
- Sant P Chawla, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maiti R. Metronomic chemotherapy. J Pharmacol Pharmacother. 2014 Jul;5(3):186-92. doi: 10.4103/0976-500X.136098. PMID 25210398
- [Background] www.accessdata.fda.gov/drugsatfda_docs (Trabectedin, Gemcitabine, Dacarbazine)